CLINICAL TRIAL: NCT00733252
Title: Optical Coherence Tomography of Human Airways
Brief Title: Optical Coherence Tomography of the Airway for Lung Cancer or Lung Disease
Status: Withdrawn | Type: Observational
Why Stopped: Low interest
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE1508; P30CA043703 (NIH); CASE1508 (Other: Case Comprehensive Cancer Center); CASE-1508-CC483
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer; Malignant Mesothelioma; Metastatic Cancer; Nonmalignant Neoplasm; Precancerous Condition
Keywords: non-small cell lung cancer; small cell lung cancer; benign respiratory tract neoplasm; lung papilloma; recurrent respiratory papillomatosis; squamous lung dysplasia; malignant mesothelioma; pulmonary carcinoid tumor; lung metastases
MeSH Terms: conditions — Lung Neoplasms; Mesothelioma, Malignant; Neoplasm Metastasis; Neoplasms; Precancerous Conditions; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Recurrent respiratory papillomatosis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Fresh Bronchi from 10 subjects undergoing pneumonectomy or lobectomy for malignant and benign processes will be obtained from the UHCMC Pathology Department as discarded tissue from fresh specimens
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: bronchoscopic and lung imaging studies — Bronchoscopic imaging and optical coherence tomography are performed on lung tissue samples collected during surgery.
Procedure: diagnostic bronchoscopy — Bronchoscopic imaging and optical coherence tomography are performed on lung tissue samples collected during surgery.
Procedure: histopathologic examination — All imaged areas are marked. The marked areas are then excised and fixed in formalin for histopathologic analysis.
Procedure: optical coherence tomography — Bronchoscopic imaging and optical coherence tomography are performed on lung tissue samples collected during surgery.

SUMMARY:
RATIONALE: Diagnostic procedures, such as optical coherence tomography, may help find and diagnose lung cancer or precancerous cells.

PURPOSE: This phase I trial is studying how well optical coherence tomography of the airway works in detecting abnormal cells in patients undergoing surgery for lung cancer or lung disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate optical coherence tomography images of the airway with airway histology.
* Develop an imaging technique to detect premalignant airway epithelial changes (carcinoma in situ, dysplasia) to study the transformation process as well as intervene and prevent the development of lung cancer.

OUTLINE: Bronchoscopic imaging and optical coherence tomography are performed on lung tissue samples collected during surgery. All imaged areas are marked. The marked areas are then excised and fixed in formalin for histopathologic analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing pneumonectomy or lobectomy for malignant or benign lung processes

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Correlation of optical coherence tomography images of the airway with airway histology | This study will involve discarded tissue from 10 subjects with pathology specimens over one year.

CONTACTS AND LOCATIONS:
Overall Officials: Rana Hejal, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://clinicaltrials.gov/ct2/show/NCT00733252?term=case1508&rank=1